CLINICAL TRIAL: NCT03751917
Title: A Long-Term Retrospective and Prospective Safety Study of Arsenic Trioxide in Patients With Newly Diagnosed, Low- to Intermediate-Risk Acute Promyelocytic Leukemia (APL)
Brief Title: Long-term Safety Study of Arsenic Trioxide in Newly Diagnosed, Low-to-intermediate Risk Acute Promyelocytic Leukemia
Acronym: APL0618
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: APL0618
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: Acute promyelocytic leukemia; Adults; Arsenic trioxide
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Arsenic Trioxide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- APL patients: The study will be conducted using multinational data from disease registries for APL. The study participants will consist of patients with newly diagnosed, low-to intermediate-risk APL.
  Interventions: Drug: Arsenic Trioxide

INTERVENTIONS:
Drug: Arsenic Trioxide — This is an observational study. Patients who have received or are receiving all trans retinoic acid (ATRA) + Arsenic Trioxide will be followed and analyzed.
  Other Names: ATRA+ATO

SUMMARY:
The therapeutic advantage of the association of ATRA + Arsenic Trioxide is more favorable and manageable as compared to ATRA + chemotherapy. Nevertheless, at present, there is not enough information on the incidence of long-term side effects.

This study, as well as other similar studies conducted around Europe, will focus on following patients treated with this therapy on a long-term basis.

Once all studies in Europe will be concluded, all data will be analyzed together.

DETAILED DESCRIPTION:
Considering the clear therapeutic advantage associated with ATRA+ATO combination therapy and the more favorable and overall manageable safety profile compared to ATRA+chemotherapy, the benefits of the combination in the first-line indication do appear to overweigh the risks.

However, no information regarding the actual adverse event (AE) incidence and the long-term toxicity of ATRA+ATO is available at present and therefore, as a postmarketing commitment, TEVA (the Company holding the Marketing Authorisation of Trisenox® (Arsenic trioxide)) is setting up a long-term safety cohort study of Trisenox in newly diagnosed low- to intermediate-risk APL patients retrospectively analyzing data from APL disease registries all around Europe.

As a result, this observational study is part of the retrospective PASS Study (A Post-Authorisation Long-Term Retrospective Safety Cohort Study of Arsenic Trioxide in First Line Low-to Intermediate-Risk Acute Promyelocytic Leukaemia Patients) that will use data from multinational APL disease registries in Europe. The present study will focus on Italian patients.

ELIGIBILITY:
Inclusion Criteria:

* APL diagnosis based on cytological criteria and confirmed by the presence of the (15;17) translocation and/or the presence of the PML/RARA rearrangement (with the determination of the breakpoint subtype).
* Newly diagnosed low- to intermediate-risk APL (white blood cells [WBC] count ≤10x103/µL)
* First line treatment with ATRA+ATO
* Aged 18 years or above
* Signed informed consent, if applicable

Exclusion Criteria:

* High risk APL (WBC count > 10x103/µL)
* APL relapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Source Population for the study is patients included in existing multinational disease registries for APL in Europe. APL registries collect real-world data on APL demographics and provide information on disease characteristics, treatment patterns and long-term effects. Participating physicians are not subject to any instructions with regard to the diagnosis and therapy of their patients. All patient treatment is carried out within routine clinical practice at the discretion of the physician and according to existing treatment guidelines.
  Data will be extracted from the registries for all patients meeting the above inclusion and exclusion criteria to provide the study population.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of grade III/IV (Common Terminology Criteria for Adverse Events (CTCAE) v4.03) adverse events of special interest (AESI). | At a maximum of 5 years from study entry
  AESI are, among others: differentiation syndrome, creatinine, bilirubin, neurotoxicity, aspartate amino transferase/alanine amino transferase (ASAT/ALAT) ratio, haemorrhage, sepsis, QTc prolongation, cardiac events including congestive heart failure (CHF).

SECONDARY OUTCOMES:
Number of unexpected serious adverse events (SAEs). | At a maximum of 5 years from study entry
  Including grading and relationship as documented in the study.
Number of patients developing secondary malignancies. | At a maximum of 5 years from study entry
Number of patients developing therapy-related myelodysplastic syndrome (tMDS). | At a maximum of 5 years from study entry
Number of patients developing acute myeloid leukemia (tAML). | At a maximum of 5 years from study entry
Number of patients who die. | At a maximum of 5 years from study entry

CONTACTS AND LOCATIONS:
Locations (28):
- Italy (28):
  - Aon Ss. Antonio E Biagio E C. Arrigo - Alessandria - Soc Ematologia, Alessandria
  - Aou Consorziale Policlinico - Bari - Uo Ematologia Con Trapianto, Bari
  - UO Ematologia con trapianto-Universita' degli Studi di Bari Aldo Moro, Bari
  - Azienda Ospedaliera - Papa Giovanni XXIII, Bergamo
  - Asst Degli Spedali Civili Di Brescia - Uo Ematologia, Brescia
  - Ao Brotzu, Presidio Ospedaliero A. Businco - Cagliari - Sc Ematologia E Ctmo, Cagliari
  - CTMO - Ematologia - Ospedale "Binaghi", Cagliari
  - U.O.C. Oncoematologia - Istituto Oncologico Veneto Irccs, Presidio Ospedaliero S. Giacomo Apostolo, Castelfranco Veneto
  - A.O. Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - U.O. di Ematologia, Catanzaro
  - Irccs Aou San Martino - Genova - Uo Ematologia E Trapianti, Genova
  - U.O.C. di Ematologia 1 e 2 IRCCS AOU San Martino-IST, Genova
  - Fondazione IRCCS Ca' Granda Osp. Maggiore Policlinico UOC Oncoematologia, Milan
  - Irccs Ospedale S. Raffaele - Milano - Uo Oncoematologia, Milan
  - Ospedale Niguarda " Ca Granda" - SC Ematologia, Milan
  - Azienda Ospedaliera "S.Gerardo", Monza
  - Napoli Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Naples
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Aou Policlinico Tor Vergata - Roma - Uoc Trapianto Cellule Staminali, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs - Roma - Area Ematologica, Roma
  - Universita' "Sapienza" - Dip Biotecnologie Cellulari - Divisione di Ematologia, Roma
  - Universita' Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Università Degli Studi Di Roma "Sapienza" - Dipartimento Di Medicina Traslazionale E Di Precisione - U.O.C. Ematologia, Roma
  - Ente Ecclesiastico Casa Sollievo Della Sofferenza - San Giovanni Rotondo - Ematologia, San Giovanni Rotondo
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia 2, Torino
  - Dipartimento di Oncologia Ematologia 2 A.O. Citta' della Salute S. G. Battista, Torino
  - Aulss 8 Berica - Ospedale Di Vicenza - Uoc Ematologia, Vicenza
  - ULSS N.6 Osp. S. Bortolo, Vicenza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: GIMEMA Foundation website — http://www.gimema.it